CLINICAL TRIAL: NCT03776266
Title: The Five-year Pattern of Red Blood Cell Transfusion and Clinical Outcome in Patients Undergoing Percutaneous Coronary Intervention: A Korean Nationwide Longitudinal Cohort Study
Brief Title: The Long-term Clinical Outcomes and Patterns of Transfusion in PCI Patients: Retrospective Cohort Study
Acronym: TFPCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Ho Choi, MD, PhD, Professor, Samsung Medical Center
Other Study IDs: SMC 2018-10-044
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Erythrocyte Transfusion; Percutaneous Coronary Intervention; Revascularization
Keywords: Transfusion; PCI; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: No intervention is required due to retrospective observational study — Red blood cell transfusion on or after percutaneous coronary intervention
  Other Names: Observation on Red blood cell transfusion on or after percutaneous coronary intervention

SUMMARY:
A nationwide retrospective cohort study. To investigate the long-term patterns of transfusion and clinical outcomes of patients undergoing PCI.

DETAILED DESCRIPTION:
A nationwide retrospective cohort study. Transfusion after PCI may increase a risk, but the long term effects after red blood cell transfusion is known. Longitudinal data is collected from administrative claims in the National Healthcare Insurance Service of Korea. All Korean patient date undergoing PCI inserting stent from January 1, 2011 to December 31, 2011 is extracted. Clinical outcomes until December 31, 2016 is investigated.

Primary outcome is the incidence density of red blood cell transfusion. Secondary outcomes are the association of transfusion with major adverse clinical event (MACE) consisting all-cause death, revascularization, critically ill cardiovascular status, or stroke.

Incidence density and time-dependent Cox proportional hazard regression is statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All Korean patients undergoing PCI using stent from January 1, 2011 to December 31, 2011

Exclusion Criteria:

* Patients without any stent insertion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing PCI using stent in 2011 from all medical providers in Korea is selected using National Healthcare Insurance System
Sampling Method: Non-Probability Sample
Enrollment: 48786 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence density of transfusion | 5 years
  5-year incidence density of red blood cell transfusion

SECONDARY OUTCOMES:
Incidence density of MACE | 5 years
  5-year incidence densities of a major adverse clinical event (MACE) consisting of all-cause death, revascularization, critically ill cardiovascular status, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ho Choi, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gang nam-Gu, Ilwon-Dong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided